CLINICAL TRIAL: NCT06846385
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II/III Seamless Clinical Study Evaluating the Efficacy, Safety, PK, PD, and ADA of MG-K10 Humanized Monoclonal Antibody Injection in the Treatment of Seasonal Allergic Rhinitis
Brief Title: Phase II/III Seamless Clinical Study of MG-K10 Humanized Monoclonal Antibody Injection in Treatment of Seasonal Allergic Rhinitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MG-K10-SAR-001
Record Dates: First submitted 2025-02-10; First posted 2025-02-26 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-02

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MG-K10 Humanized Monoclonal Antibody Injection (Experimental): A single dose was administered
  Interventions: Biological: MG-K10 Humanized Monoclonal Antibody Injection
- placebo (Placebo Comparator): A single dose was administered
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — A single dose was administered
  Arms: placebo
Biological: MG-K10 Humanized Monoclonal Antibody Injection — MG-K10 Humanized Monoclonal Antibody Injection
  Arms: MG-K10 Humanized Monoclonal Antibody Injection

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled Phase II/III seamless clinical study evaluating the efficacy, safety, pharmacokinetic (PK) profile, pharmacodynamic (PD) profile, and immunogenicity of MG-K10 humanized monoclonal antibody injection in the treatment of seasonal allergic rhinitis

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo-controlled Phase II/III seamless clinical study evaluating the efficacy, safety, pharmacokinetic (PK) profile, pharmacodynamic (PD) profile, and immunogenicity of MG-K10 humanized monoclonal antibody injection in the treatment of seasonal allergic rhinitis.

About 120 patients with seasonal allergic rhinitis in stage II and 106 patients with monthly seasonal allergic rhinitis in stage III received only one dose. The study was divided into a screening period (1 week), a double-blind treatment period (4 weeks) and a safety follow-up period (2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-75 years old (including the cutoff value), male or female;
* With reference to the diagnosis and treatment of allergic rhinitis China guide (2022 revision) "subjects conforms to the diagnosis of seasonal allergic rhinitis, history 2 years or more clear, at the same time, at least one over the same period of the current season or allergic rhinitis disease related Skin prick test (Skin Prick Test, SPT) or serum Specific IgE (sIgE) (acceptable within less than 1 year before randomization), and the results met the diagnostic criteria for SAR
* During the previous pollen season, the subjects used nasal corticosteroids or other SAR drugs (antihistamines, leukotriene receptor antagonists, etc.), and their SAR symptoms were poorly controlled.
* The following criteria were met at screening and baseline:

  1. iTNSS score at screening ≥6, nasal congestion ≥2, runny nose, nasal itching, and sneezing 3. One of the symptoms ≥2 points;
  2. iTNSS score ≥6 at baseline; rTNSS≥6 points, nasal congestion ≥2 points, runny nose, nose,one of the three symptoms of itching and sneezing ≥2 points
* Throughout the study period (from signing the ICF to 6 months after the study drug administration), fertile female subjects and their partners agreed to use highly effective birth control, and male subjects and their partners agreed to use effective birth control and had no plans to donate sperm (men) or eggs (women)
* Be able to understand and comply with clinical protocol requirements, voluntarily participate in clinical trials, and subjects voluntarily sign written informed consent.

Exclusion Criteria:

* Allergy to the study drug or its excipients;
* Travel plans for 48 hours or more from known pollen areas during the screening/induction and treatment periods (visit 5);
* The subject's exposure to allergens in his or her home or work environment may have changed significantly during the trial, which the investigator determines may affect the efficacy evaluator;
* Subjects with limited outdoor activities during the day were defined as those who did not have any outdoor activities during the day for 1 or 4 days per week.

  ·Patients who have previously received anti-interleukin-4 receptor alpha (IL-4Rα) monoclonal antibody drugs (such as dupriuzumab) for Allergic Rhinitis (AR) have poor response (such as treatment failure or treatment intolerance);
* Use of antihistamines within 4 days prior to randomization;
* Leukotriene receptor antagonists and hypertrophic cell membrane stabilizers were used within 1 week before randomization;
* Received medium - and short-acting Systemic Crticosteroids (SCS, including oral, intravenous and intramuscular glucocorticoids) and Chinese medicine for AR treatment (systemic Chinese medicine preparation) within 4 weeks before randomization. Had received long-acting SCS (such as triamcinolone olone injection) within 6 weeks prior to randomization, or planned to receive these medications during the study period;
* Participants with asthma who began inhaled glucocorticoid therapy within the first 4 weeks of randomization.
* Stable dose inhaled glucocorticoids were used for at least 4 weeks and evaluated before randomization
* The dose of inhaled glucocorticoids was maintained during the study period, while the dosage of inhaled glucocorticoids was ≤1000 μg/ day of fluticasone propionate or equivalent doses of other inhaled glucocorticoids
* Randomized 8 weeks or 5 Systemic immunosuppressants (including but not limited to methotrexate, cyclosporine, mycophenolate, tacrolimus, penicillamine, sulfasulazopyridine, hydroxychloroquine, azathioprine, cyclophosphamide) have been used within a half-life (whichever is longer) to treat inflammatory or autoimmune diseases (e.g., rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic disease) Lupus erythematosus, multiple sclerosis, etc);
* random or 10 weeks before 5 within the half-life of longer (in time) received anti IL - 4 r alpha monoclonal antibody, Thymic Stromal lymphocytes (Thymic Stromal Lymphopoietin, TSLP) monoclonal antibody, anti-IGE monoclonal antibody, other monoclonal antibody or other biologic agent therapy;
* Participated in MG-K10 clinical trials;
* Live/attenuated vaccine received within 3 months prior to randomization or during the planned study period; Subjects who started Immunotherapy [including Intravenous Immunoglobin (IVIG) therapy or Specific Immunotherapy (SIT) therapy] within 6 months before randomization, Participants who plan to begin immunotherapy during the study;
* Had received any nasal or sinus surgery within 1 year prior to randomization;
* History of vital organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation
* Other nasal comorbiditis or co-occurring diseases/conditions (such as acute/chronic sinusitis, nasal polyps, deviation of nasal septum, drug-induced rhinitis, cerebrospinal fluid rhinorrhea, nasal postoperative status within 1 year, etc.) were present at the time of screening and could affect the efficacy evaluation as assessed by the investigators;
* Acute sinusitis, nasal infection, or upper respiratory tract infection during the screening/induction period or within 2 weeks prior to screening;
* Have malignant or benign tumors in the nasal cavity;
* Screening for infections requiring treatment with systemic antimicrobials, antivirals, antifungals, antiparasites or antigenics within 7 days prior to the visit;
* Patients with Perennial Allergic Rhinitis (PAR) who are allergic to pet hair (if the subject is currently free of pet hair contact) may be included. PAR subjects who are allergic to other indoor allergens may be included);
* Have a history of lymphoproliferative diseases, or have had or are present with malignant tumors within 5 years prior to screening (except for skin squamous cell carcinoma in situ, basal cell carcinoma, and cervical carcinoma in situ after thorough treatment without any signs of recurrence);
* Have a history or evidence of high risk cardiovascular disease
* Have posterior subcapsular cataracts or glaucoma, or any other eye condition that may affect the evaluation of eye symptoms, or related conditions listed below
* Active TB infection is present or suspected;
* Presence or suspected worm infection within 6 months;
* A history of severe herpes virus infection, such as herpes encephalitis, disseminated herpes, etc.
* Patients with severe diseases of the central nervous system, respiratory system, liver, kidney, gastrointestinal, urinary, endocrine, or blood systems that the investigator believes may affect the efficacy and safety of the subject;
* Known or suspected immunosuppressed individuals, including, but not limited to, a history of invasive opportunistic infections (e.g., tuberculosis, histoplasmosis, listeriosis, coccidioidosis, pulmonary cyst disease, aspergillosis), even if the infection has resolved; Or unusual frequent, recurrent, or long-term infections (as determined by the investigator)
* The presence of any significant laboratory anomalies
* Pregnant or lactating women, or those with a positive pre-randomized serum pregnancy test
* According to the judgment of the researcher, it is not suitable to participate in this researcher for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean rTNSS from baseline after 2 weeks of treatment | 2 weeks

SECONDARY OUTCOMES:
Rate of change of mean rTNSS from baseline after 2 weeks of treatment | 2 weeks
Rate of change of mean rTNSS from baseline after 4 weeks of treatment | 4 weeks
Change in mean instantaneous total nasal symptom score from baseline after 2 and 4 weeks of treatment | 2 and 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No